CLINICAL TRIAL: NCT05238064
Title: PI3Kδ Inhibitor Parsaclisib in Combination With Cyclophosphamide, Doxorubicin, Vincristine and Prednisone in Participants With Previously Untreated Peripheral T-cell Lymphoma
Brief Title: Parsaclisib in Combination With CHOP in Participants With Previously Untreated PTCL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Junning Cao, MD, Vice dean of department of oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTCL-2022-01
Record Dates: First submitted 2022-01-28; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: PI3Kδ Inhibitor; Parsaclisib; CHOP; PTCL
MeSH Terms: interventions — parsaclisib; Cyclophosphamide; Doxorubicin; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PI3Kδ inhibitor Parsaclisib plus CHOP (Experimental): Phase Ib (Explored the appropriate dose of Parsaclisib in combination with CHOP)
  Parsaclisib is taken orally every day continuously, at approximately the same time every day, without food restriction, once a day.
  CHOP was given at the standard dose, 21 days per cycle
  Phase II:
  Induced treatment: Received the initial dose of Parsaclisib determined in Phase Ib day 1-14 of each cycle, as well as CHOP at standard dose for 6 cycles.
  Maintain treatment: Parsaclisib maintenance (2.5mg po, qd) will be performed on CR or PR patients after 6 cycles of induction therapy until disease progression, death, unacceptable toxicity, withdrawal of informed consent, or the investigator's decision or initiation of new antitumor therapy. The maximum maintenance period of parsaclisib is 24 months.
  Interventions: Drug: Parsaclisib; Drug: CHOP

INTERVENTIONS:
Drug: Parsaclisib — Phase Ib: Parsaclisib is taken orally every day continuously, at approximately the same time every day, without food restriction, once a day. This stage follows the traditional "3+3" model. Parsaclisib is set at 10 mg/day, 15 mg/day, 20 mg/day 3 dose groups, starting from 10 mg/day, each group included 3 subjects. The final dose determined at this stage will be used in the Phase II study.
  Phase II:
  Induced treatment: Received the initial dose of Parsaclisib determined in Phase Ib.
  Maintain treatment: 2.5mg orally every day continuously, once a day until disease progression, death or unacceptable toxicity developments. The maximum treatment time of Parsaclisib is no more than 2 years.
  Other Names: IBI376
Drug: CHOP — Cyclophosphamide: 750mg/m2, IV, d1 Doxorubicin: 50mg/m2, IV, d1 Vincristine: 1.4mg/m2, IV, d1 (maximum 2mg) Prednison: 100mg, po, d1-5 21 days per cycle
  Other Names: Cyclophosphamide, doxorubicin, vincristine and prednison

SUMMARY:
The study is to investigate the safety, tolerability and efficacy of PI3Kδ inhibitor Parsaclisib in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) in frontline treatment of patients with peripheral T-cell lymphoma (PTCL).

DETAILED DESCRIPTION:
The study is to investigate the safety, tolerability and efficacy of PI3Kδ inhibitor Parsaclisib in combination with cyclophosphamide, doxorubicin, vincristine and prednisone (CHOP) in frontline treatment of patients with peripheral T-cell lymphoma (PTCL) by conducting in two stages, dose-escalation stage and dose-expansion stage. In dose-escalation stage, patients with treated-naïve PTCL will be assigned to receive sequentially higher doses of parsaclisib range from 10 to 20mg po, qd plus CHOP (21 days per cycle). The dose escalation will follow the classic 3+3 design. The recommended phase 2 dose (RP2D) of parsaclisib will be determined according to the dose-escalation results. In dose-expansion stage, additional patients will be recruited to receive Par-CHOP for the planned 6 cycles or until disease progression, unacceptable drug-related adverse events or starting new anti-lymphoma treatments.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects fully understand and voluntarily participate in this study and sign informed consent
* 2. Age≥18, ≤70 years
* 3. Histologically confirmed diagnosis of treatment-naïve PTCL, including peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), anaplastic large cell lymphoma (ALCL, ALK+ALCL with IPI≥2, no limitation with ALC-ALCL), angioimmunoblastic T-cell lymphoma (AITL), enteropathy related T-cell lymphoma, hepatosplenic T-cell, γ/δ T-cell lymphoma; Other PTCL that investigators consider to be appropriate to be enrolled.
* 4. No previous systemic treatment before enrollment.
* 5. At least one measurable lesions according to LUGANO 2014 criteria.
* 6. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-2.
* 7. Life expectancy ≥3 months.
* 8. Ineligible or decline to receive autologous stem cell transplantation (ASCT).
* 9. Adequate main organ function defined as the following required baseline laboratory data: Absolute neutrophil count (ANC)≥1.5×109/L without given G-CSF within 14 days; Platelet count (PLT)≥75×109/L without given transfusion with 14 days; Hemoglobin (HB)≥8g/dL without given transfusion or erythropoietin; Total bilirubin (TBIL)≤1.5X upper limit of normal (ULN); Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5X ULN; Serum creatinine (Scr)≤1.5X ULN; Left ventricular ejection fraction (LVEF)≥50%; For female participants of childbearing period, a negative urine or serum pregnancy test should be performed with 1 week prior to receiving first dose of investigational drug (day 1 of cycle 1). If a urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required. Women of non-reproductive age was defined as at least 1 year after menopause or having undergone surgical sterilization or hysterectomy.
* 10.If there is a risk of pregnancy, all participants (both men and women) are required to use a contraceptive with an annual failure rate of less than 1% for entire treatment period up to 120 days after the last dose of investigational drug (or 180 days after chemotherapeutic drug).

Exclusion Criteria:

* 1. Current or previous history of other malignancies within 5 years prior to study enrollment.
* 2. Current diagnosis of any of the following: Adult T-cell leukemia/lymphoma, precursor cell lymphoblastic leukemia/lymphoma, extranodal natural killer/T-cell lymphoma, nasal type (ENKTL), indolent cutaneous T-cell lymphoma (CTCL).
* 3. Target lesions were treated with radiotherapy within 4 weeks of enrollment.
* 4. Patients undergo interventional clinical trials.
* 5. Concurrent lymphoma with CNS invasion.
* 6. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation.
* 7. Known allergy to the active ingredients or excipients of IBI376 and CHOP regimens.
* 8. A known history of human immunodeficiency virus (HIV) infection (i.e., HIV antibody positive).
* 9. Positive test results for HBsAg antigen and HBV-DNA, or hepatitis C virus (HCV) antibody.
* 10. Received live vaccine within 30 days prior to initial investigational drug administration (day 1 of cycle 1) (Note: inactivated virus vaccine for injection is allowed within 30 days prior to initial administration, but live attenuated vaccine is not allowed).
* 11. Pregnant or breastfeeding women.
* 12. Any serious uncontrolled systemic disease.
* 13. Any medical history or disease evidence that may interfere with the study results or other conditions that investigators consider inappropriate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
3-year EFS | From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  the period from the date of patients sign informed consent to the observed progression of the disease or the occurrence of death for any reason

SECONDARY OUTCOMES:
Hematology and non hematology toxicity | Throughout the treatment period，up to 6 months
  number of participants with treatment-related adverse events as assessed by CTCAE v5.0
CRR | at the end of Cycle 6 (each cycle is 21 days)
  the ratio of numbers of patients with complete response to all the participants receiving treatment
ORR | at the end of Cycle 6 (each cycle is 21 days)
  the ratio of numbers of patients with complete response and partial response to all the participants receiving treatment
EFS | From date of randomization until the date of first documented event, such as progression of the disease or the occurrence of death for any reason, or receive other anti-tumor treatment, whichever came first, assessed up to 3 years
  the period from the date of patients sign informed consent to the observed event, such as progression of the disease or the occurrence of death for any reason, or receive other anti-tumor treatment
OS | From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 3 years
  time between the date of patients sign informed consent and the date of death or the date of last follow-up time

CONTACTS AND LOCATIONS:
Overall Officials: Junning Cao, Principal Investigator — Fudan University